CLINICAL TRIAL: NCT03503838
Title: A Pilot Study of Online Yoga to Improve Symptom Burden (i.e., Fatigue) and Quality of Life in MPN Patients
Brief Title: A Pilot Study of Online Yoga for MPN Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004303
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Quality of Life; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention group with a wait-list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Yoga (Experimental): The intervention will be 12 weeks in duration and will consist of a series of pre-approved online yoga classes. MPN patients will be asked to complete a minimum of 60 minutes per week of yoga practice with encouragement to do more if they can. All Udaya.com videos will include a proper warm-up, cool down, and closing mindfulness activity (i.e., message from yoga therapist, brief meditation, final relaxation). Qualified Udaya yoga instructors who collectively have over 200 years of training and experience will expertly instruct the online yoga classes.
  Interventions: Behavioral: Online Yoga
- Wait-List Control (No Intervention): The control group will be asked to maintain their usual level of activity for 16 weeks before being given access to the yoga intervention. Once study participants in the yoga group have completed all outcome measures up through the 4-week follow-up (week 16), participants in the control group will be allowed to participate in the same online yoga prescription that was provided to the yoga group.

INTERVENTIONS:
Behavioral: Online Yoga — 12 weeks of online yoga; 60 min/week
  Arms: Online Yoga

SUMMARY:
Polycythemia vera (PV), essential thrombocytosis (ET), and myelofibrosis (MF) are chronic Philadelphia negative myeloproliferative neoplasms (MPNs) that are characterized by clonal proliferation of hematopoietic stem cells, intramedullary fibrosis, and splenomegaly. While disease manifestations may vary amongst the spectrum of MPNs, quality of life considerations including fatigue, concentration difficulties, pain, sleep disturbance, and depression are negatively affected in most MPN patients. Inflammation has been suggested to be involved in the development of disease-related symptoms. Specific pro-inflammatory cytokines (e.g., IL-1, IL-6, IL-8, and TNF-α) have been associated with particular patient-reported symptoms, including fatigue, abdominal complaints, microvascular symptoms, and constitutional symptoms. Pharmacologic therapy can positively impact MPN related symptoms, specifically with JAK inhibition, however, these treatments often come with negative side effects (e.g., anemia, thrombocytopenia). Much opportunity remains for improving MPN symptoms (i.e., fatigue, insomnia, loss of muscle mass, and debilitation) and quality of life.

Yoga, a gentle form of meditative exercise, has been shown to improve symptom management and quality of life parameters in cancer patients and may be effective in improving MPN-related symptoms. Here we propose a study evaluating the efficacy of an online yoga intervention comparing a yoga group to a wait-list control group for improving symptom burden and quality of life in MPN patients. Secondarily, we plan to evaluate the feasibility of collecting potential biomarkers that are related to MPN disease-related activity, such as fatigue (i.e., cortisol and serum cytokines).

DETAILED DESCRIPTION:
Participants will be recruited nationally utilizing internet-based strategies, including social media (i.e., Facebook, Twitter), social networking sites, online and email listervs, and by contacting MPN patients that were not included in prior feasibility work but expressed their interest in future work. The research team will provide flyers to recruitment contacts to provide a description of the study.

MPN patients that expressed interest in future studies will be contacted via email to be asked of their interest in the current study. A flyer will be provided in the email. Prospective organizations will be contacted via email and/or phone and asked to advertise the study by posting the provided recruitment information (e.g., flyers, blurbs) to social media sites and/or websites, emailing listservs, or displaying flyers at location. National organizations agreeing to advertise for the study will be sent recruitment information (e.g., flyers, blurbs) via email, and local organizations will have the option for hand delivery or email. Interested MPN patients will complete an eligibility screening using a Qualtrics link. The eligibility screening takes 5-10 minutes to complete.

If ineligible, the participant will be sent an email notification and will be offered a discounted monthly membership to online yoga streaming (Udaya.com). If eligible, the potential participant will be emailed to schedule a time for an intake appointment. The intake appointment will provide greater details pertaining to the study, review of the consent process, and address participant questions.

After completing the intake appointment, the participant will be directed to an informed consent page (individual link using Qualtrics) with details concerning the requirements of the study, as well as potential risks and benefits. There will be a place for the participant to type in their electronic signature, which will constitute their consent to participate in the study. After receipt of the signed consent form, the participant will be mailed a Fitbit. They will be instructed to wear the Fitbit for one week to collect baseline physical activity. After one week of wear, the participant will be directed to a Qualtrics link to complete baseline self-report measures. At this point, the participant will be randomized into either the wait-list control group or the yoga group via a web-based randomization tool.

Yoga Group: The intervention will be 12-weeks in duration and will consist of a series of pre-approved online yoga classes. MPN patients will be asked to complete a minimum of 60 minutes per week of yoga practice with encouragement to do more if they can. All Udaya.com videos will include a proper warm-up, cool down, and closing mindfulness activity (i.e., message from yoga therapist, brief meditation, final relaxation). A 12-week yoga prescription utilized in prior feasibility work will be improved and modified for this study. The 12-week yoga prescription was designed to be safe and progressive for this specific population. Modifications to the prescription will be made based on qualitative feedback received from patients that participated in prior feasibility work. During the intervention, all classes will offer alternative poses, modifications, and use of props (i.e., yoga blocks and straps) in the instance poses are difficult for the participant (i.e., painful, irregular, uneven breath) and to ensure safety. In addition to specific instruction regarding form and safety, the yoga therapist will provide descriptions of each video that includes tips and modifications to poses (e.g., set the knee on your yoga mat if this feels more comfortable for you). Additionally, patients will also receive a yoga modifications handout outlining the contraindicated yoga poses with modifications. This handout will include an exercise warning for patients that experience dizziness, lightheadedness or faintness, excessive shortness of breath, chest pain, and that they need to stop the activity and contact their health care professional immediately if these symptoms are experienced.

Wait-List Control Group: The control group will be asked to maintain their usual level of activity for 16 weeks before being given access to the yoga intervention. Once study participants in the yoga group have completed all outcome measures up through the 4-week follow-up (week 16), participants in the control group will be allowed to participate in the same online yoga prescription that was provided to the yoga group.

ELIGIBILITY:
Inclusion Criteria:

1) have a diagnosis of essential thrombocytosis, polycythemia vera, or myelofibrosis identified by treating physician, 2) answer "no" to all items on the Physical Activity Readiness Questionnaire (PAR-Q), or be willing to obtain a signed medical release from their physician in the case that a question is answered with a "yes", 3) have access to a desktop or laptop on a regular basis, 4) have access to reliable internet, 5) read and understand English, 6) age 18 years or older, 7) willing to be randomized to a yoga group or a wait-list control group, and 8) willing to drive to the nearest Patient Service Center in order to receive a blood draw

Exclusion Criteria:

1) Currently perform Tai Chi, Qi Gong, or Yoga at least 60 min or more weekly, 2) currently engage in ≥150 min/week of moderate-/vigorous-intensity physical activity on a weekly basis, 3) have a history of syncope in last 2 months, 4) have a history of recurrent falls (≥2 in 2 months), 5) have a score of ≥15 on the Patient Health Questionnaire 9 (PHQ-9) indicating moderate-severe levels of depression, 6) have an Eastern Cooperative Oncology Group 3 (ECOG 3) questionnaire score greater than three, 7) currently utilize Udaya.com, 8) currently pregnant, or 9) currently reside outside of the United States of America

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Symptom Burden | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  A 10-item, validated form that calculates total symptom burden score (MPN Symptom Assessment Form Total Symptom Score)
Change in Fatigue | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  A single-item fatigue question taken from the MPN Symptom Assessment Form
Change in Anxiety | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  NIH PROMIS Anxiety Short Form
Change in Depression | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  NIH PROMIS Depression Adult Short Form
Change in Sleep Disturbance | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  NIH PROMIS Sleep Disturbance Adult Short Form
Change in Sexual Function | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  NIH PROMIS Sexual Function
Change in Pain Intensity | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  NIH PROMIS Pain Intensity Adult Short Form
Change in Global Health | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  NIH PROMIS Global Health

SECONDARY OUTCOMES:
Change in Inflammatory Cytokine Profile | Change from baseline to week 12 and change from baseline to week 16 (follow-up)
  IL-6, TNF-a as measured in blood samples from study participants

IPD SHARING:
Plan to Share IPD: Undecided
De-identified participant data will be shared with researchers upon reasonable request.

REFERENCES:
- [Derived] Huberty J, Eckert R, Dueck A, Kosiorek H, Larkey L, Gowin K, Mesa R. Online yoga in myeloproliferative neoplasm patients: results of a randomized pilot trial to inform future research. BMC Complement Altern Med. 2019 Jun 7;19(1):121. doi: 10.1186/s12906-019-2530-8. PMID 31174535